### Permission to Take Part in a Human Research Study



#### **University at Buffalo Institutional Review Board (UBIRB)**

Office of Research Compliance | Clinical and Translational Research Center Room 5018 875 Ellicott St. | Buffalo, NY 14203 UB Federalwide Assurance ID#: FWA00008824

**Title of research study:** Developing health information interventions 3

Version Date: 1/28/25

Investigator: Heather Orom, PhD

**<u>Key Information</u>**: The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

#### Why am I being invited to take part in a research study?

You are being invited to take part in a research study to help develop new ways of communicating about health.

#### What should I know about a research study?

- This information sheet will explain the study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.

# Why is this research being done?

We are conducting this research in order to develop innovative ways of communicating about cancer prevention.

## How long will the research last and what will I need to do?

We expect that participating in the study will take 9 minutes. You will be asked to watch a video and answer survey questions about your personal characteristics, feelings and behavior. You will also be invited to take part in a very brief (about 2 minutes) survey nine months from now in which you will be asked to answer a few questions about your behavior.

## Is there any way being in this study could be bad for me?

We do not anticipate that there is any way being in the study could be bad for you.

## Will being in this study help me in any way?

There are no benefits to you from your taking part in this research. We cannot promise any benefits to others from your taking part in this research. However, possible benefits to others include improved ways of reaching people with cancer information.

HRPP Revision Date: Jan 11, 2019 Page 1 of 2

## Permission to Take Part in a Human Research Study

### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You may choose not to enroll in this study. You may choose to withdraw from the study at any time. Your alternative to participating in this research study is to not participate.

#### How many people will be studied?

We expect about 1,500 people will be in this study.

#### What happens if I say yes, but I change my mind later?

You can leave the research at any time it will not be held against you. You may contact IPSOS to have your data removed from the study.

## What happens to the information collected for the research?

Only anonymous data will be shared with the researchers.

#### Who is paying for this research?

This research is being funded by the National Institutes of Health

#### Will I get paid for my participation in this research?

You will receive your standard incentive.

#### What will happen to my information?

Your information may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

Your study information will not be used for future studies and no identifying information is collected for this project.

If you have questions, concerns, or complaints, or think the research has hurt you, you may also talk to the research team at horom@buffalo.edu or 716-829-6682; however, in this case your participation in the study may no longer be anonymous. You may also contact the research participant advocate at 716-888-4845 or researchadvocate@buffalo.edu.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). An IRB is a committee that provides ethical and regulatory oversight of research that involves human subjects. You may talk to them at (716) 888-4888 or email ub-irb@buffalo.edu if:

- You have questions about your rights as a participant in this research
- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You want to get information or provide input about this research.

## Would you like to participate in this research?

By advancing to the survey you are indicating your willingness to participate in the research.

HRPP Revision Date: Jan 11, 2019 Page 2 of 2